CLINICAL TRIAL: NCT05542290
Title: Implantation of Capsular Tension Ring in Primary Angle Closure Patients With Zonular Laxity or Dialysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Principal Investigator, Chunyan Qiao_2021, Ophthalmologist, Professor, M.D., Beijing Tongren Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BeijingTH-CTR
Record Dates: First submitted 2022-09-03; First posted 2022-09-15 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Glaucoma; Angle-Closure
Keywords: angle closure; zonular laxity; zonular dialysis; lens subluxation; capsular tension ring; efficacy; safety
MeSH Terms: conditions — Glaucoma; Lens Subluxation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With capsular tension ring implantation (Experimental): We performed phacoemulsification lens extraction and intraocular lens implantation with capsular tension ring implantation combined with goniosynechialysis.
  Interventions: Procedure: Capsular tension ring implantation
- Without capsular tension ring implantation (Other): We performed phacoemulsification lens extraction and intraocular lens implantation without capsular tension ring implantation combined with goniosynechialysis.
  Interventions: Procedure: No capsular tension ring implantation

INTERVENTIONS:
Procedure: Capsular tension ring implantation — Capsular tension ring implantation during phacoemulsification lens extraction and intraocular lens implantation combined with goniosynechialysis in included angle closure patients.
  Arms: With capsular tension ring implantation
Procedure: No capsular tension ring implantation — No capsular tension ring implantation during phacoemulsification lens extraction and intraocular lens implantation combined with goniosynechialysis in included angle closure patients.
  Arms: Without capsular tension ring implantation

SUMMARY:
Primary angle closure glaucoma (PACG) is the main type of glaucoma in China, which includes acute and chronic PACG. According to the International Society of Geographical and Epidemiological Ophthalmology (ISGEO), this spectrum of disease is divided into acute angle closure crisis (AACC), primary angle closure suspect (PACS), primary angle closure (PAC) and PACG. Previous researchers have reported that with the wider use of lens extraction and intraocular lens (IOL) implantation combined with anti-glaucoma surgery in the treatment of PAC and PACG, the prevalence of zonular laxity or dialysis in primary angle closure disease (PACD) was found to be relatively high. In one of the studies performed by the investigators, the proportion of zonular laxity or dialysis was 46.2%, significantly higher than that in the age-related cataract patients (control group), which was 6.0%. In PACD patients with zonular laxity or dialysis, whether or not should the investigators implant capsular tension ring (CTR), the efficacy and safety of CTR implantation, and if there is any difference in the prevalence of complications during and after surgery between patients with and without CTR implantation remain unclear. The purpose of this study was to investigate the efficacy and safety of CTR implantation in PACD patients with zonular laxity and zonular dialysis ≤ 4 clocks.

DETAILED DESCRIPTION:
Patients with PACD who are scheduled to have phacoemulsification and IOL implantation combined with goniosynechialysis are recruited. All recruited patients attended comprehensive eye examinations and interviews. Past history of ocular and systemic diseases, family and personal history, history of ocular trauma and surgery were interviewed. And the patients underwent ophthalmic examinations including visual acuity tests (presenting visual acuity [PVA] and best-corrected visual acuity [BCVA]), subjective refraction, intraocular pressure (IOP) measurements, slit-lamp examination, fundus photography, gonioscopy, ocular biometry using IOL Master 700, ultrasound biomicroscopy, anterior segment optical coherence tomography (ASOCT) imaging. All patients provide informed consent for inclusion in the study.

All surgery procedures were performed by the same surgeons (CYQ) using the same standard operation procedure. All patients use the same type of foldable IOL calculated using SRK/T formula. During the surgery, patients with wrinkling of the anterior capsule (multiple sinusoidal folds were formed) during continuous curvilineal capsulorhexis (CCC) at the needle or forceps tip but without infolding of peripheral capsule or visualisation of the capsular equator during the cortical or nuclear removal, or, wrinkling of the anterior capsule during CCC with infolding of peripheral capsule and visualisation of the capsular equator ≤ 4 clocks of range during the cortical or nuclear removal, were finally included in the study and randomly assigned (using a random-number table generated by SAS) with equal probability to either CTR group (with CTR implantation during the surgery) and control group (without CTR implantation during the surgery). All patients included in the CTR group use the same type of CTR. The investigators recorded the complications during the surgery including vitreous prolapse, hyphema, vitreous hemorrhage, damage of iris and lens capsule, et al.

Postoperatively, all patients received similar routine medication comprising topical prednisolone acetate (six times a day for 1 week and tapered down by 1 time every week), topical levofloxacin hydrochloride (four times a day for 1 month), and Tobramycin and Dexamethasone Eye Ointment (1 time every night for 1 month).

Postoperative examinations were performed at 1 day, 1 week, 1 months, 3 months, 6 months and 12 months. During the follow-up visits, a complete ophthalmic examination was performed including PVA, BCVA, subjective refraction, non-contact IOP measurement, slit-lamp examination, slit-lamp photography after pupil dilation, ASOCT, gonioscopy, and fundus imaging.

ELIGIBILITY:
Inclusion Criteria:

* Age: 45-79 years old
* Continuous cases diagnosed with AACC, PACS, PAC and PACG in glaucoma department of Beijing Tongren Hospital from October 1st, 2022 to December 31th, 2024 and undergo phacoemulsification lens extraction and intraocular lens implantation combined with goniosynechialysis
* Wrinkling of the anterior capsule during manual continuous circular capsulorhexis (CCC) but without infolding of peripheral capsule or visualization of the capsular equator, or, wrinkling of the anterior capsule during manual capsulorhexis and combined with visualization of capsular equator and infolding of peripheral capsule ≤ 4 clocks (lens subluxation)
* The eye of each subject that meet the inclusion criteria is included and if both eyes meet the inclusion criteria, the first eye that undergo the surgery is included

Exclusion Criteria:

* Past history of intraocular surgeries including trabeculectomy, peripheral iridotomy, glaucoma valve implantation, vitrectomy, and so on
* Past history of laser peripheral iridotomy or iridoplasty
* Past history of ocular trauma or signs referring to ocular trauma
* Ocular diseases that may cause zonulopathy, including choroidal detachment, retinal detachment, ciliary body detachment, intraocular tumor and so on
* Lens related secondary glaucoma, including spherophakia, Marfan syndrome, homocystinuria and son on
* Other secondary angle closure glaucoma, including neovascular glaucoma, iritis related secondary glaucoma and so on
* Visualization of capsular equator and infolding of peripheral capsule > 4 clocks during the surgery
* Anterior or posterior capsule rupture during the surgery which makes it impossible for CTR implantation

Ages: 45 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Spherical equivalent | baseline
  Sphere +1/2 cylinder obtained from subjective refraction
Spherical equivalent | 1 month after the surgery
  Sphere +1/2 cylinder obtained from subjective refraction
Spherical equivalent | 3 months after the surgery
  Sphere +1/2 cylinder obtained from subjective refraction
Spherical equivalent | 6 months after the surgery
  Sphere +1/2 cylinder obtained from subjective refraction
Spherical equivalent | 12 months after the surgery
  Sphere +1/2 cylinder obtained from subjective refraction
Area of anterior capsulorhexis | 1 week after the surgery
  Area of anterior capsulorhexis measured using slit-lamp photography
Area of anterior capsulorhexis | 1 month after the surgery
  Area of anterior capsulorhexis measured using slit-lamp photography
Area of anterior capsulorhexis | 3 months after the surgery
  Area of anterior capsulorhexis measured using slit-lamp photography
Area of anterior capsulorhexis | 6 months after the surgery
  Area of anterior capsulorhexis measured using slit-lamp photography
Area of anterior capsulorhexis | 12 months after the surgery
  Area of anterior capsulorhexis measured using slit-lamp photography
Assessment of posterior capsular opacification | 1 week after the surgery
  Assessment of posterior capsular opacification using slit-lamp photography
Assessment of posterior capsular opacification | 1 month after the surgery
  Assessment of posterior capsular opacification using slit-lamp photography
Assessment of posterior capsular opacification | 3 months after the surgery
  Assessment of posterior capsular opacification using slit-lamp photography
Assessment of posterior capsular opacification | 6 months after the surgery
  Assessment of posterior capsular opacification using slit-lamp photography
Assessment of posterior capsular opacification | 12 months after the surgery
  Assessment of posterior capsular opacification using slit-lamp photography
The extent of iris-trabecular contact | baseline
  The extent of iris-trabecular contact assessed by gonioscopy
The extent of iris-trabecular contact | 1 month after the surgery
  The extent of iris-trabecular contact assessed by gonioscopy
The extent of iris-trabecular contact | 3 months after the surgery
  The extent of iris-trabecular contact assessed by gonioscopy
The extent of iris-trabecular contact | 6 months after the surgery
  The extent of iris-trabecular contact assessed by gonioscopy
The extent of iris-trabecular contact | 12 months after the surgery
  The extent of iris-trabecular contact assessed by gonioscopy
The extent of peripheral anterior synechia | baseline
  The extent of peripheral anterior synechia assessed by gonioscopy
The extent of peripheral anterior synechia | 1 month after the surgery
  The extent of peripheral anterior synechia assessed by gonioscopy
The extent of peripheral anterior synechia | 3 months after the surgery
  The extent of peripheral anterior synechia assessed by gonioscopy
The extent of peripheral anterior synechia | 6 months after the surgery
  The extent of peripheral anterior synechia assessed by gonioscopy
The extent of peripheral anterior synechia | 12 months after the surgery
  The extent of peripheral anterior synechia assessed by gonioscopy
Corneal thickness | baseline
  Corneal thickness obtained by IOL Master 700
Central anterior chamber depth | baseline
  Central anterior chamber depth obtained by IOL Master 700
Lens thickness | baseline
  Lens thickness obtained by IOL Master 700
Axial Length | baseline
  Axial Length obtained by IOL Master 700
Refractive prediction error | baseline
  Refractive prediction error obtained by IOL Master 700
Anterior chamber depth | baseline
  Anterior chamber depth obtained by anterior segment optical coherence tomography
Anterior chamber depth | 1 week after the surgery
  Anterior chamber depth obtained by anterior segment optical coherence tomography
Anterior chamber depth | 1 month after the surgery
  Anterior chamber depth obtained by anterior segment optical coherence tomography
Anterior chamber depth | 3 months after the surgery
  Anterior chamber depth obtained by anterior segment optical coherence tomography
Anterior chamber depth | 6 months after the surgery
  Anterior chamber depth obtained by anterior segment optical coherence tomography
Anterior chamber depth | 12 months after the surgery
  Anterior chamber depth obtained by anterior segment optical coherence tomography
Angle opening distance | baseline
  Angle opening distance obtained by anterior segment optical coherence tomography
Angle opening distance | 1 week after the surgery
  Angle opening distance obtained by anterior segment optical coherence tomography
Angle opening distance | 1 month after the surgery
  Angle opening distance obtained by anterior segment optical coherence tomography
Angle opening distance | 3 months after the surgery
  Angle opening distance obtained by anterior segment optical coherence tomography
Angle opening distance | 6 months after the surgery
  Angle opening distance obtained by anterior segment optical coherence tomography
Angle opening distance | 12 months after the surgery
  Angle opening distance obtained by anterior segment optical coherence tomography
Trabecular-iris space area | baseline
  Trabecular-iris space area obtained by anterior segment optical coherence tomography
Trabecular-iris space area | 1 week after the surgery
  Trabecular-iris space area obtained by anterior segment optical coherence tomography
Trabecular-iris space area | 1 month after the surgery
  Trabecular-iris space area obtained by anterior segment optical coherence tomography
Trabecular-iris space area | 3 months after the surgery
  Trabecular-iris space area obtained by anterior segment optical coherence tomography
Trabecular-iris space area | 6 months after the surgery
  Trabecular-iris space area obtained by anterior segment optical coherence tomography
Trabecular-iris space area | 12 months after the surgery
  Trabecular-iris space area obtained by anterior segment optical coherence tomography
Trabecular-iris angle | baseline
  Trabecular-iris angle obtained by anterior segment optical coherence tomography
Trabecular-iris angle | 1 week after the surgery
  Trabecular-iris angle obtained by anterior segment optical coherence tomography
Trabecular-iris angle | 1 month after the surgery
  Trabecular-iris angle obtained by anterior segment optical coherence tomography
Trabecular-iris angle | 3 months after the surgery
  Trabecular-iris angle obtained by anterior segment optical coherence tomography
Trabecular-iris angle | 6 months after the surgery
  Trabecular-iris angle obtained by anterior segment optical coherence tomography
Trabecular-iris angle | 12 months after the surgery
  Trabecular-iris angle obtained by anterior segment optical coherence tomography
Anterior chamber width | baseline
  Anterior chamber width obtained by anterior segment optical coherence tomography
Anterior chamber width | 1 week after the surgery
  Anterior chamber width obtained by anterior segment optical coherence tomography
Anterior chamber width | 1 month after the surgery
  Anterior chamber width obtained by anterior segment optical coherence tomography
Anterior chamber width | 3 months after the surgery
  Anterior chamber width obtained by anterior segment optical coherence tomography
Anterior chamber width | 6 months after the surgery
  Anterior chamber width obtained by anterior segment optical coherence tomography
Anterior chamber width | 12 months after the surgery
  Anterior chamber width obtained by anterior segment optical coherence tomography
Iris thickness | baseline
  Iris thickness obtained by anterior segment optical coherence tomography
Iris thickness | 1 week after the surgery
  Iris thickness obtained by anterior segment optical coherence tomography
Iris thickness | 1 month after the surgery
  Iris thickness obtained by anterior segment optical coherence tomography
Iris thickness | 3 months after the surgery
  Iris thickness obtained by anterior segment optical coherence tomography
Iris thickness | 6 months after the surgery
  Iris thickness obtained by anterior segment optical coherence tomography
Iris thickness | 12 months after the surgery
  Iris thickness obtained by anterior segment optical coherence tomography
Iris cross-sectional area | baseline
  Iris cross-sectional area obtained by anterior segment optical coherence tomography
Iris cross-sectional area | 1 week after the surgery
  Iris cross-sectional area obtained by anterior segment optical coherence tomography
Iris cross-sectional area | 1 month after the surgery
  Iris cross-sectional area obtained by anterior segment optical coherence tomography
Iris cross-sectional area | 3 months after the surgery
  Iris cross-sectional area obtained by anterior segment optical coherence tomography
Iris cross-sectional area | 6 months after the surgery
  Iris cross-sectional area obtained by anterior segment optical coherence tomography
Iris cross-sectional area | 12 months after the surgery
  Iris cross-sectional area obtained by anterior segment optical coherence tomography
Iris curvature | baseline
  Iris curvature obtained by anterior segment optical coherence tomography
Iris curvature | 1 week after the surgery
  Iris curvature obtained by anterior segment optical coherence tomography
Iris curvature | 1 month after the surgery
  Iris curvature obtained by anterior segment optical coherence tomography
Iris curvature | 3 months after the surgery
  Iris curvature obtained by anterior segment optical coherence tomography
Iris curvature | 6 months after the surgery
  Iris curvature obtained by anterior segment optical coherence tomography
Iris curvature | 12 months after the surgery
  Iris curvature obtained by anterior segment optical coherence tomography
Lens thickness | baseline
  Lens thickness obtained by anterior segment optical coherence tomography
Lens thickness | 1 week after the surgery
  Lens thickness obtained by anterior segment optical coherence tomography
Lens thickness | 1 month after the surgery
  Lens thickness obtained by anterior segment optical coherence tomography
Lens thickness | 3 months after the surgery
  Lens thickness obtained by anterior segment optical coherence tomography
Lens thickness | 6 months after the surgery
  Lens thickness obtained by anterior segment optical coherence tomography
Lens thickness | 12 months after the surgery
  Lens thickness obtained by anterior segment optical coherence tomography
Lens vault | baseline
  Lens vault obtained by anterior segment optical coherence tomography
Lens vault | 1 week after the surgery
  Lens vault obtained by anterior segment optical coherence tomography
Lens vault | 1 month after the surgery
  Lens vault obtained by anterior segment optical coherence tomography
Lens vault | 3 months after the surgery
  Lens vault obtained by anterior segment optical coherence tomography
Lens vault | 6 months after the surgery
  Lens vault obtained by anterior segment optical coherence tomography
Lens vault | 12 months after the surgery
  Lens vault obtained by anterior segment optical coherence tomography
The distance between intraocular lens and the posterior capsular | 1 week after the surgery
  The distance between intraocular lens and the posterior capsular obtained by CASIA2 anterior segment optical coherence tomography
The distance between intraocular lens and the posterior capsular | 1 month after the surgery
  The distance between intraocular lens and the posterior capsular obtained by CASIA2 anterior segment optical coherence tomography
The distance between intraocular lens and the posterior capsular | 3 months after the surgery
  The distance between intraocular lens and the posterior capsular obtained by CASIA2 anterior segment optical coherence tomography
The distance between intraocular lens and the posterior capsular | 6 months after the surgery
  The distance between intraocular lens and the posterior capsular obtained by CASIA2 anterior segment optical coherence tomography
The distance between intraocular lens and the posterior capsular | 12 months after the surgery
  The distance between intraocular lens and the posterior capsular obtained by CASIA2 anterior segment optical coherence tomography
Intraocular lens inclination angle | 1 week after the surgery
  Intraocular lens inclination angle obtained by CASIA2 anterior segment optical coherence tomography
Intraocular lens inclination angle | 1 month after the surgery
  Intraocular lens inclination angle obtained by CASIA2 anterior segment optical coherence tomography
Intraocular lens inclination angle | 3 months after the surgery
  Intraocular lens inclination angle obtained by CASIA2 anterior segment optical coherence tomography
Intraocular lens inclination angle | 6 months after the surgery
  Intraocular lens inclination angle obtained by CASIA2 anterior segment optical coherence tomography
Intraocular lens inclination angle | 12 months after the surgery
  Intraocular lens inclination angle obtained by CASIA2 anterior segment optical coherence tomography
Effective intraocular lens position | 1 week after the surgery
  Effective intraocular lens position obtained by CASIA2 anterior segment optical coherence tomography
Effective intraocular lens position | 1 month after the surgery
  Effective intraocular lens position obtained by CASIA2 anterior segment optical coherence tomography
Effective intraocular lens position | 3 months after the surgery
  Effective intraocular lens position obtained by CASIA2 anterior segment optical coherence tomography
Effective intraocular lens position | 6 months after the surgery
  Effective intraocular lens position obtained by CASIA2 anterior segment optical coherence tomography
Effective intraocular lens position | 12 months after the surgery
  Effective intraocular lens position obtained by CASIA2 anterior segment optical coherence tomography
The distance between ciliary body and the equator of lens at 3 o'clock position | baseline
  The distance between ciliary body and the equator of lens at 3 o'clock position obtained by ultrasound biomicroscopy
The distance between ciliary body and the equator of lens at 6 o'clock position | baseline
  The distance between ciliary body and the equator of lens at 6 o'clock position obtained by ultrasound biomicroscopy
The distance between ciliary body and the equator of lens at 9 o'clock position | baseline
  The distance between ciliary body and the equator of lens at 9 o'clock position obtained by ultrasound biomicroscopy
The distance between ciliary body and the equator of lens at 12 o'clock position | baseline
  The distance between ciliary body and the equator of lens at 12 o'clock position obtained by ultrasound biomicroscopy
Incidence of complications | 1 month after the surgery
  Incidence of complications including posterior capsular opacification (PCO), IOL tilt, capsule contraction syndrome, et al.
Incidence of complications | 3 months after the surgery
  Incidence of complications including PCO, IOL tilt, capsule contraction syndrome, et al.
Incidence of complications | 6 months after the surgery
  Incidence of complications including PCO, IOL tilt, capsule contraction syndrome, et al.
Incidence of complications | 12 months after the surgery
  Incidence of complications including PCO, IOL tilt, capsule contraction syndrome, et al.

SECONDARY OUTCOMES:
Presenting visual acuity | baseline
  Presenting visual acuity with or without glasses
Presenting visual acuity | 1 day after the surgery
  Presenting visual acuity with or without glasses
Presenting visual acuity | 1 week after the surgery
  Presenting visual acuity with or without glasses
Presenting visual acuity | 1 month after the surgery
  Presenting visual acuity with or without glasses
Presenting visual acuity | 3 months after the surgery
  Presenting visual acuity with or without glasses
Presenting visual acuity | 6 months after the surgery
  Presenting visual acuity with or without glasses
Presenting visual acuity | 12 months after the surgery
  Presenting visual acuity with or without glasses
Best corrected visual acuity | baseline
  Visual acuity with refractive correction
Best corrected visual acuity | 1 month after the surgery
  Visual acuity with refractive correction
Best corrected visual acuity | 3 months after the surgery
  Visual acuity with refractive correction
Best corrected visual acuity | 6 months after the surgery
  Visual acuity with refractive correction
Best corrected visual acuity | 12 months after the surgery
  Visual acuity with refractive correction
Intraocular pressure | baseline
  Intraocular pressure obtained by non-contact tonometer
Intraocular pressure | 1 day after the surgery
  Intraocular pressure obtained by non-contact tonometer
Intraocular pressure | 1 week after the surgery
  Intraocular pressure obtained by non-contact tonometer
Intraocular pressure | 1 month after the surgery
  Intraocular pressure obtained by non-contact tonometer
Intraocular pressure | 3 months after the surgery
  Intraocular pressure obtained by non-contact tonometer
Intraocular pressure | 6 months after the surgery
  Intraocular pressure obtained by non-contact tonometer
Intraocular pressure | 12 months after the surgery
  Intraocular pressure obtained by non-contact tonometer
Number of anti-glaucoma medications | 1 week after the surgery
  Number of anti-glaucoma medications
Number of anti-glaucoma medications | 1 month after the surgery
  Number of anti-glaucoma medications
Number of anti-glaucoma medications | 3 months after the surgery
  Number of anti-glaucoma medications
Number of anti-glaucoma medications | 6 months after the surgery
  Number of anti-glaucoma medications
Number of anti-glaucoma medications | 12 months after the surgery
  Number of anti-glaucoma medications
Vertical cup-to-disc ratio | baseline
  Vertical cup-to-disc ratio evaluated by fundus photography
Vertical cup-to-disc ratio | 1 month after the surgery
  Vertical cup-to-disc ratio evaluated by fundus photography
Vertical cup-to-disc ratio | 6 months after the surgery
  Vertical cup-to-disc ratio evaluated by fundus photography
Vertical cup-to-disc ratio | 12 months after the surgery
  Vertical cup-to-disc ratio evaluated by fundus photography

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tongren Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No